CLINICAL TRIAL: NCT06786039
Title: Clinical Impact of Non-invasive Neurally Adjusted Ventilatory Assist in Very Preterm Infants
Status: Recruiting | Type: Observational
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Juyoung Lee, Professor, Korea University Anam Hospital
Other Study IDs: 2024AN0554
Record Dates: First submitted 2025-01-06; First posted 2025-01-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Preterm Infant
Keywords: infant, premature; Noninvasive NAVA
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NIV-NAVA application: Preterm infants born between 27 weeks 0 days to 31 weeks 6 days of gestation requiring respiratory support within 48 hours after birth
  Interventions: Procedure: Non-invasive NAVA

INTERVENTIONS:
Procedure: Non-invasive NAVA — Initiate respiratory assist with NIV-NAVA within 48 hours. The setting of respiratory support will be adjusted based on clinical conditions of each subject. NIV-NAVA could be switched to nasal continuous airway pressure or high flow nasal cannula, and it also could be stopped after initial stabilization.
  In cases of respiratory distress syndrome, lung surfactant will be administered via the less invasive surfactant administration (LISA) method and avoid endotracheal intubation whenever possible. For who intubated in the delivery room, extubation with NIV-NAVA should be considered as soon as possible. Endotracheal intubation with invasive ventilation could be applied when clinical deteriorations happens.

SUMMARY:
This is a prospective observational study investigating the impact of NIV-NAVA on short-term clinical outcomes and long-term neurodevelopment in very preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 27 weeks 0 days to 31 weeks 6 days of gestation
* Preterm infants who require respiratory support within the first 48 hours of life

Exclusion Criteria:

* Preterm infants who die within the first 48 hours of life
* Preterm infants who do not require any respiratory support within the first 48 hours of life.
* Preterm infants with congenital anomalies affecting the lungs, heart, or other organs that could influence breathing
* Infants whose parents do not consent to participate in the study

Ages: 1 Hour to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients admitted to the NICU in Korea University Anam Hospital will be recruited over a 2-year period.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2029-12-20 (Estimated); Study Completion 2030-12-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Non-invasive neurally adjusted ventilatory assist (NIV-NAVA) failure | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  NIV-NAVA failure was defined as a participant requiring endotracheal intubation (except brief intubation for only surfactant administration)

SECONDARY OUTCOMES:
Rate of bronchopulmonary dysplasia (BPD) | at 36 weeks of postmenstrual age
  diagnosed according to the Jensen Criteria
Duration of non-invasive ventilation | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  each of NIV-NAVA, nasal continuous positive airway pressure, high flow nasal cannula
Incidence of periventricular leukomalacia (PVL) | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  diagnosed by brain ultrasound or MRI
Duration of invasive ventilation | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  each of high-frequent oscillatory ventilation, conventional mechanical ventilation, NAVA etc
Incidence of air leaks | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  including pneumothorax, pneumomediastinum and pulmonary interstitial emphysema
Incidence of patent ductus arteriosus (PDA) | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  defined by clinical and/or echocardiographic criteria requiring symptomatic treatment (except prophylaxis)
Time to achieve full enteral feeding | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  day of life when milk amount reaches 100 mL/kg/day or higher
Incidence of intraventricular hemorrhage (IVH) | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  defined by the Papile criteria, using cranial ultrasonography (≥grade 2)
Incidence of retinopathy of prematurity (ROP) | through the study completion, during the hospital stay in neonatal intensive care unit up to 3 months
  defined according to the international classification of ROP (≥stage 2)
Total brain volume (mL) | term equivalent age defined as 37-42 weeks mean postmenstrual age at brain MRI
  Total brain volume (TBV) will be measured from Brain MRI
Intracranial volume (mL) | term equivalent age defined as 37-42 weeks mean postmenstrual age at brain MRI
  Intracranial volume (ICV) will be measured from Brain MRI
Relative sizes of volumes of particular regions of interest | term equivalent age defined as 37-42 weeks mean postmenstrual age at brain MRI
  relative sizes of volumes of particular regions of interest (ROIs) will be measured from brain MRI
Bayley Scales of Infant Development III - 2 yr | 18-24 months of corrected age
  scale scores for each development areas (cognitive, language, motor) score range : 0-200 above average (1-2 SD, score 116-130) average ( 1 to 1 SD, score 85-115) below average (1 to-2 SD, score 84-70) well below average (<-2 SD, scores < 70).
Modified Checklist for Autism in Toddlers (M-CHAT) | 18-24 months of corrected age
  autism spectrum disorder screening test result total score 0-2: low risk total score 3-7: moderate risk total score 8-20: high risk
MacArthur-Bates Communication Development Inventory | 18-24 months of corrected age
  language evaluation questionnaire result The criterion for identifying risk for delayed language development was an expressive vocabulary size <10th percentile
Bayley Scales of Infant Development III - 3 yr | 33-39 months of age
  scale scores for each development areas (cognitive, language, motor) score range : 0-200 above average (1-2 SD, score 116-130) average ( 1 to 1 SD, score 85-115) below average (1 to-2 SD, score 84-70) well below average (<-2 SD, scores < 70).
Child Behavior Checklist (CBCL) | 33-39 months of age
  behavior screening questionnaire result t-score ≤ 59: non-clinical symptoms, t-score between 60 and 64: at risk for problem behaviors t-score ≥ 65: clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National Bundang Hospital NICU, Seongnam-si, Gyeonggi-do
  - Korea University Anam Hospital, NICU, Seoul

IPD SHARING:
Plan to Share IPD: Undecided